CLINICAL TRIAL: NCT01463839
Title: Association Between Quality of Sleep and Harmful Oral Habits Among Children
Brief Title: Sleep Disorder and Oral Habits in Children
Acronym: SOHab
Status: Completed | Type: Observational
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Lara Jansiski Motta, PhD, University of Nove de Julho
Other Study IDs: hab026/2010
Record Dates: First submitted 2011-10-28; First posted 2011-11-02 (Estimated); Last update posted 2011-11-02 (Estimated); Status verified 2011-10

CONDITIONS: Sleep Disorder; Malocclusion
Keywords: sleep disorder; malocclusion; children
MeSH Terms: conditions — Sleep Wake Disorders; Malocclusion

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Children 3 to 6: Fifty children (3 to 6 years of age) from a private school in the city of Sao Paulo

SUMMARY:
Sleep is a vital physiological function for the maintenance of health and quality of life. Harmful, non-nutritive and parafunctional oral habits are believed to have a negative effect on adequate rest at night. The aim of the present study was to determine associations between quality of sleep and harmful oral habits among children aged three to six years. Fifty children from a private school in São Paulo (Brazil) were evaluated using two questionnaires on sleep quality and harmful oral habits. The data were submitted to descriptive analysis. The chi-square test was employed for the categorical variables and analysis of variance (ANOVA) was carried out to compare mean values. The Student's t-test was used for all analyses, with the significance level set at 5%. The SPSS 12.0 program for Windows was used to analyze the results.

DETAILED DESCRIPTION:
An observational cross-sectional study was carried out with the aim of determining associations between quality of sleep and harmful oral habits among children aged three to six years. This study was conducted in compliance with the Brazilian National Health Council/Ministry of Health guidelines contained in Resolution 196/96 and received approval from the Human Research Ethics Committee of the Universidade Metropolitana de Santos (Brazil) under process number 026/2010. Parents/guardians of all participants were properly informed regarding the objectives of the study and signed a statement of informed consent.

Fifty children (3 to 6 years of age) from a private school in the city of Sao Paulo were evaluated by means of two questionnaires administered to parents/guardians: The "Undesirable Habits Questionnaire", composed of 15 investigative questions on harmful oral habits as well as dietary and psychological factors, and the Sleep Habits Questionnaire.6 The data were submitted to descriptive analysis. The chi-square test was employed for the categorical variables and analysis of variance (ANOVA) was carried out to compare mean values. The Student's t-test was used for all analyses, with the significance level set at 5%. The SPSS 12.0 program for Windows was used to analyze the results.

ELIGIBILITY:
Inclusion Criteria:

* 3 to 6 years of age

Exclusion Criteria:

* over 6 years of age

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Fifty children (3 to 6 years of age) from a private school in the city of Sao Paulo
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2010-09; Primary Completion 2010-10 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lara Motta, PhD, Principal Investigator — Nove de Julho University
Locations (1):
- Nove de Julho University, São Paulo, São Paulo, Brazil